CLINICAL TRIAL: NCT01333189
Title: Improving Function After Knee Arthroplasty With Weight-Bearing Biofeedback
Acronym: RELOAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 10-1185; 2558404 (Other: unknwn); K23AG029978 (NIH); R01HD065900 (NIH); T32AG000279 (NIH)
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Arthropathy of Knee Joint
Keywords: total knee arthroplasty; osteoarthritis; biomechanics; gait
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RELOAD: Weight-bearing biofeedback exercise (Experimental): RELOAD participants participated in two 30-minute training sessions/week with a physical therapist for a total of 6 weeks, focusing on promoting WB symmetry using a progressive series of activities adapted to video games. These biofeedback training sessions were provided in addition to the standard of care rehabilitation that the CONTROL group received. Total dose of exercise across groups was matched.
  Interventions: Other: Weight-bearing biofeedback exercise
- CONTROL: Standard of care exercise (Active Comparator): CONTROL participants were provided two weeks of home rehabilitation (6 visits) by a physical therapist. Patients then progressed to outpatient rehabilitation, consisting of 4 weeks of treatment for a total of 6 weeks of standard of care rehabilitation. Total dose of exercise across groups was matched.
  Interventions: Other: Standard of care exercise

INTERVENTIONS:
Other: Weight-bearing biofeedback exercise — Patients in the experimental group completed the same standard of care rehabilitation program as the control group. Thus, the experimental intervention was in addition to the standard intervention.
  Upon discharge to home, patients in the RELOAD group began the weight bearing (WB) biofeedback phase of the study. Patients participated in two 30-minute training sessions/week with a physical therapist for a total of 6 weeks, focusing on promoting WB symmetry using a progressive series of activities adapted to video games.
  Arms: RELOAD: Weight-bearing biofeedback exercise
Other: Standard of care exercise — Standard inpatient rehabilitation began on post-operative day 1 and lasted for an average of 3.2 days. After hospital discharge, two weeks of home rehabilitation (6 visits) were provided by physical therapists. Patients progressed to outpatient rehabilitation, consisting of 4 weeks of treatment. As such, 6 weeks of rehabilitation following hospital discharge was implemented for both groups.
  Arms: CONTROL: Standard of care exercise

SUMMARY:
The purpose of this study is to determine if rehabilitation using weight-bearing biofeedback training following total knee arthroplasty (TKA) is more effective than standard rehabilitation methods in promoting weight-bearing symmetry through the lower limbs during functional activities such as sit-to-stand transfers and walking. Secondary outcomes of interest include functional measures and internal moment at the hip, knee, and ankle joints during sit-to-stand and walking.

DETAILED DESCRIPTION:
People who have had knee replacement surgery typically have worse physical function compared to healthy people of similar age. This problem occurs despite completion of standard rehabilitation programs. One reason for less-than-optimal restoration of physical function is that standard rehabilitation does not effectively address habitual movement patterns that persist after surgery. These movement patterns are characterized by patients placing less weight on their surgical leg compared to their non-surgical leg after surgery. This asymmetrical movement pattern has been identified by researchers and shown to not completely resolve after knee replacement surgery, even though the surgery reliably reduces knee pain. The persistence of asymmetrical weight-bearing during every day activity may limit the stimulus needed for full recovery by the muscles and joints of the surgical leg. By promoting increased loading of the surgical leg, a greater stimulus can be provided to promote better functional recovery, compared with standard rehabilitation. As a result, people may subsequently move more symmetrically with improved recovery of physical function. Improved function would in turn promote the person's ability to participate in life events, limiting disability. Considering that over 500,000 knee replacement surgeries occur in the United States each year, maximizing functional recovery and limiting disability following surgery are important goals.

The investigators propose a new method of exercising following knee replacement surgery. This method involves using a commercially available game system to promote "re-loading" of the surgical limb. The game system has games designed to allow the person playing to move objects or characters on a screen by shifting his/her weight from one leg to another while standing on an instrumented "balance board". The investigators have developed an exercise program to promote shifting weight to the surgical limb, by choosing appropriate games and manipulating the goals of those games. It is the investigators' hypothesis that early application of this surgical leg "re-loading" intervention after knee replacement will result in meaningful improvement in physical function by improving movement symmetry.

ELIGIBILITY:
Inclusion Criteria:

* unilateral total knee arthroplasty, body mass index <40 kg/m^2

Exclusion Criteria:

* neurological, vascular or cardiac problems that limited physical function, contralateral knee pain greater than 2/10 on a numerical pain rating scale, severe osteoarthritis or other orthopaedic conditions in the non-operated lower extremity that limited function, sub-acute inpatient rehabilitation following unilateral total knee arthroplasty, uncontrolled diabetes, smoking or drug abuse, living >45 minutes away from the outpatient rehabilitation clinic, surgical complication requiring an altered course of rehabilitation, inability to walk 30 meters without an assistive device or inability to rise from a chair without use of arms

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory L Christiansen, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Background] Mizner RL, Snyder-Mackler L. Altered loading during walking and sit-to-stand is affected by quadriceps weakness after total knee arthroplasty. J Orthop Res. 2005 Sep;23(5):1083-90. doi: 10.1016/j.orthres.2005.01.021. Epub 2005 Mar 28. PMID 16140191
- [Background] Boonstra MC, Schwering PJ, De Waal Malefijt MC, Verdonschot N. Sit-to-stand movement as a performance-based measure for patients with total knee arthroplasty. Phys Ther. 2010 Feb;90(2):149-56. doi: 10.2522/ptj.20090119. Epub 2009 Dec 10. PMID 20007664
- [Background] Christiansen CL, Bade MJ, Judd DL, Stevens-Lapsley JE. Weight-bearing asymmetry during sit-stand transitions related to impairment and functional mobility after total knee arthroplasty. Arch Phys Med Rehabil. 2011 Oct;92(10):1624-9. doi: 10.1016/j.apmr.2011.05.010. Epub 2011 Aug 12. PMID 21839986
- [Background] Yoshida Y, Zeni J, Snyder-Mackler L. Do patients achieve normal gait patterns 3 years after total knee arthroplasty? J Orthop Sports Phys Ther. 2012 Dec;42(12):1039-49. doi: 10.2519/jospt.2012.3763. Epub 2012 Oct 22. PMID 23090437
- [Derived] Christiansen CL, Bade MJ, Davidson BS, Dayton MR, Stevens-Lapsley JE. Effects of Weight-Bearing Biofeedback Training on Functional Movement Patterns Following Total Knee Arthroplasty: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2015 Sep;45(9):647-55. doi: 10.2519/jospt.2015.5593. Epub 2015 Jul 24. PMID 26207975

RESULTS

PARTICIPANT FLOW:
Groups:
- RELOAD: Weight-bearing Biofeedback Exercise: RELOAD participants participated in two 30-minute training sessions/week with a physical therapist for a total of 6 weeks, focusing on promoting WB symmetry using a progressive series of activities adapted to video games. These biofeedback training sessions were provided in addition to the standard of care rehabilitation that the CONTROL group received. Total dose of exercise across groups was matched.
  Weight-bearing biofeedback exercise: Patients in the experimental group completed the same standard of care rehabilitation program as the control group. Thus, the experimental intervention was in addition to the standard intervention.
  Upon discharge to home, patients in the RELOAD group began the weight bearing (WB) biofeedback phase of the study. Patients participated in two 30-minute training sessions/week with a physical therapist for a total of 6 weeks, focusing on promoting WB symmetry using a progressive series of activities adapted to video games.
- CONTROL: Standard of Care Exercise: CONTROL participants were provided two weeks of home rehabilitation (6 visits) by a physical therapist. Patients then progressed to outpatient rehabilitation, consisting of 4 weeks of treatment for a total of 6 weeks of standard of care rehabilitation.
  Standard of care exercise: Standard inpatient rehabilitation began on post-operative day 1 and lasted for an average of [3] days. After hospital discharge, two weeks of home rehabilitation (6 visits) were provided by physical therapists. Patients progressed to outpatient rehabilitation, consisting of 4 weeks of treatment. As such, 6 weeks of rehabilitation following hospital discharge was implemented for both groups.
Period: Overall Study
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2
Not completed — Time constraints | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Transportation difficulties | 0 | 1
Not completed — Moved from region | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.6) | 66.6 (8.1) | 67.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Weight-bearing Ratio During Five Times Sit-to-Stand Test (FTSST)
Description: Weight-bearing ratio is measured during transitions between sitting and standing and is indicated by symmetry in vertical ground reaction force (vGRF) between lower limbs. Ratios reported are (vGRF of the Surgical Limb):(vGRF Non-Surgical Limb).
Time Frame: 6 weeks post-operative
Population: At the completion of the intervention (6 weeks post-operative), one patient from each group had dropped out of the study due to either time constraints or transportation difficulties.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
ratio | 0.77 (0.1) | 0.8 (0.11)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.329, Mixed Models Analysis

2. Secondary Outcome: Weight-bearing Ratio During Walking
Description: Weight-bearing ratio is measured during walking as the ratio between lower limbs in peak vertical ground reaction force (vGRF) during the loading response phase of the stance period of gait. Ratios reported are (vGRF of the Surgical Limb):(vGRF Non-Surgical Limb).
Time Frame: 6 weeks post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
ratio | 0.94 (0.08) | 0.92 (0.09)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.891, Mixed Models Analysis

3. Secondary Outcome: Five Times Sit-to-Stand Test (FTSST)
Description: The Five Times Sit-to-Stand Test is quantified as the total time required for an individual to rise from and return to a chair five times in a row.
Time Frame: 6 weeks post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
seconds | 11.5 (1.6) | 12.7 (3.3)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis

4. Secondary Outcome: Hip, Knee, and Ankle Joint Moments During Five Times Sit-to-Stand Test
Description: Internal joint moments at the hip, knee, and ankle were calculated using an inverse dynamics approach from data collected using embedded force plates and a 6-camera motion analysis system to assess reflective marker positions placed at landmarks of the upper limbs, trunk, and lower limbs.
Time Frame: 6 weeks post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton-meters per kilogram (Nm/kg)
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
Newton-meters per kilogram (Nm/kg)
  Hip Moment | 0.73 (0.28) | 0.80 (0.26)
  Knee Moment | 0.77 (0.21) | 0.72 (0.18)
  Ankle Moment | 0.29 (0.14) | 0.31 (0.17)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the hip; Test type: Superiority or Other; p = 0.509, Mixed Models Analysis
Statistical Analysis 2: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the knee; Test type: Superiority or Other; p = 0.500, Mixed Models Analysis
Statistical Analysis 3: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the ankle; Test type: Superiority or Other; p = 0.607, Mixed Models Analysis

5. Secondary Outcome: Walking Speed
Description: Self-selected walking speed was recorded for three passes across the middle 6 meter section of a walkway. The average of the 3 passes is reported.
Time Frame: 6 weeks post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
meters/second | 1.20 (0.23) | 1.16 (0.2)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis

6. Secondary Outcome: Hip, Knee, and Ankle Joint Moments During Walking
Description: as for outcome 4
Time Frame: 6 weeks post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton-meters per kilogram (Nm/kg)
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 12 | 12
Newton-meters per kilogram (Nm/kg)
  Hip Moment | 0.28 (0.26) | 0.26 (0.21)
  Knee Moment | 0.47 (0.22) | 0.46 (0.37)
  Ankle Moment | 0.17 (0.23) | 0.17 (0.32)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the hip; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis
Statistical Analysis 2: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the knee; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis
Statistical Analysis 3: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the ankle; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis

7. Secondary Outcome: Weight-bearing Ratio During Five Times Sit-to-Stand Test (FTSST)
Description: as for outcome 1
Time Frame: 26 weeks post-operative
Population: At the long-term follow up time point (26 weeks post-operative), a total of two patients from each group had dropped out of the study due to time constraints, transportation difficulties, late infection, or moving away from the area.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
ratio | 0.88 (0.11) | 0.91 (0.13)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.511, Mixed Models Analysis

8. Secondary Outcome: Weight-bearing Ratio During Walking
Description: as for outcome 2
Time Frame: 26 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
ratio | 0.98 (0.06) | 0.93 (0.06)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.402, Mixed Models Analysis

9. Secondary Outcome: Five Times Sit-to-Stand Test (FTSST)
Description: as for outcome 3
Time Frame: 26 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
seconds | 9.5 (2.4) | 9.6 (1.6)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis

10. Secondary Outcome: Hip, Knee, and Ankle Joint Moments During Five Times Sit-to-Stand Test
Description: as for outcome 4
Time Frame: 26 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Newton-meters per kilogram (Nm/kg)
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
Newton-meters per kilogram (Nm/kg)
  Hip Moment | 0.65 (0.24) | 0.63 (0.20)
  Knee Moment | 1.03 (0.22) | 0.97 (0.11)
  Ankle Moment | 0.17 (0.16) | 0.24 (0.14)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the hip; Test type: Superiority or Other; p = 0.686, Mixed Models Analysis
Statistical Analysis 2: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the knee; Test type: Superiority or Other; p = 0.434, Mixed Models Analysis
Statistical Analysis 3: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the ankle; Test type: Superiority or Other; p = 0.227, Mixed Models Analysis

11. Secondary Outcome: Walking Speed
Description: as for outcome 5
Time Frame: 26 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
meters/second | 1.29 (0.25) | 1.24 (0.13)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis

12. Secondary Outcome: Hip, Knee, and Ankle Moments During Walking
Description: as for outcome 4
Time Frame: 26 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Newton-meters per kilogram (Nm/kg)
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Number analyzed (Participants) | 11 | 11
Newton-meters per kilogram (Nm/kg)
  Hip Moment | 0.28 (0.19) | 0.36 (0.22)
  Knee Moment | 0.61 (0.25) | 0.42 (0.44)
  Ankle Moment | 0.09 (0.29) | 0.01 (0.19)
Statistical Analysis 1: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the hip; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis
Statistical Analysis 2: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the knee; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis
Statistical Analysis 3: Comparison: RELOAD: Weight-bearing Biofeedback Exercise vs CONTROL: Standard of Care Exercise; Internal moment at the ankle; Test type: Superiority or Other; p = 0.877, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 26 weeks following total knee arthroplasty (TKA)
Arm/Group | RELOAD: Weight-bearing Biofeedback Exercise | CONTROL: Standard of Care Exercise
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RELOAD: Weight-bearing Biofeedback Exercise (N=13) | CONTROL: Standard of Care Exercise (N=13)
Late Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes